CLINICAL TRIAL: NCT00127842
Title: Rating Evaluations in Psoriatic Arthritis (PsA) With Enbrel®
Brief Title: REPArE: Rating Evaluations in Psoriatic Arthritis (PsA) With Etanercept (Enbrel®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040131
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; PsA; Commercial product; American College of Rheumatology; ACR/PASI
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Etanercept

ARMS (1):
- Etanercept (Other): Open-label etanercept administered by subcutaneous injection at a dose of 50 mg/week for 24 months.
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Administered according to the product monograph by subcutaneous (SC) injection
  Other Names: Enbrel®

SUMMARY:
The overall objective of the study was to describe the long-term effectiveness and safety of etanercept in patients with psoriatic arthritis in a Canadian clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* Presence of psoriasis or previous evidence of psoriasis documented by a dermatologist as part of usual care
* At least one of the following forms of psoriatic arthritis (PsA):

  * Distal interphalangeal (DIP) involvement (inflammatory)
  * Polyarticular arthritis, absence of rheumatoid nodules and presence of psoriasis
  * Arthritis mutilans
  * Asymmetric peripheral arthritis or
  * Spinal involvement
* Active psoriatic arthritis at the time of the study enrollment
* Patients must demonstrate greater than 3 swollen joints and greater than 3 tender/painful joints
* Greater than 18 years of age at the time of consent
* Able to start etanercept therapy per the approved product monograph
* Informed consent must be provided before any study specific procedures are performed

Exclusion Criteria:

* Active infections at time of initiating Enbrel® therapy
* Evidence of skin conditions (e.g., eczema) other than psoriasis that would interfere with evaluations of the study medication
* A malignancy, other than basal cell carcinoma of the skin or, in situ carcinoma of the cervix, within the past 5 years
* Known hypersensitivity to etanercept or any of its components
* Patients receiving, or who have received:

  * Remicade® (infliximab) in the previous 3 months or -- Humira® (adalimumab) in the previous 3 months or
  * Kineret® (anakinra) in the previous 15 days
* Patients receiving or who have received etanercept
* Treatment with any investigational therapy in the 30 days prior to enrollment or during the study
* Active guttate, erythrodermic or pustular psoriasis at the time of screening
* Presence of any significant and uncontrolled medical condition, which in the Investigator's opinion, precludes the use of etanercept as outlined in the product monograph
* Sepsis or at risk of septic syndrome
* Patients not available for follow-up assessment
* Concerns for subject's compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-08; Primary Completion 2005-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Gladman DD, Bombardier C, Thorne C, Haraoui B, Khraishi M, Rahman P, Bensen W, Syrotuik J, Poulin-Costello M. Effectiveness and safety of etanercept in patients with psoriatic arthritis in a Canadian clinical practice setting: the REPArE trial. J Rheumatol. 2011 Jul;38(7):1355-62. doi: 10.3899/jrheum.100698. Epub 2011 May 15. PMID 21572156
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 5 August 2005 through 2 February 2007
Groups:
- Enbrel: Open-label etanercept administered by subcutaneous injection at a dose of 50 mg/week for 24 months.
Period: Overall Study
Arm/Group | Enbrel
Started | 110
Completed | 71
Not Completed | 39
Not completed — Adverse Event | 15
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 12
Not completed — Noncompliance | 2
Not completed — Protocol Violation | 1
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Enbrel
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 54
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 1
  Chinese | 1
  Other Asian | 2
  Canadian Aboriginal | 2
  Other | 1
  Caucasian | 103
Health and Labour Questionnaire (HLQ) Absence from Work Module [Mean (Standard Deviation); unit: days] — The HLQ collects quantitative data on the relation between illness and treatment and work performance. The instrument is divided into 4 modules to collect data about absence from work, reduced productivity at paid work, unpaid labor production and impediments to paid and unpaid labor. The absence from work module asks participants to indicate how many days in the past 2 weeks they missed work due to health problems.
  days | 0.8 (2.51)
HLQ Reduced Productivity at Paid Work Module [Mean (Standard Deviation); unit: Hours] — The reduced productivity at work module of the HLQ asks participants to estimate the number of additional hours required to compensate for production losses due to illness on working days over the past 2 weeks.
  Hours | 2.3 (8.22)
HLQ Unpaid Work Module: Help Received with Unpaid Work [Mean (Standard Deviation); unit: Hours] — The Unpaid Labour Production Module of the HLQ assesses the amount of hours of unpaid work (including household work, shopping, caring for children and odd jobs around the house), normally performed by the participant, that were taken over by other members of the household, family or friends (unpaid help), and/or by paid workers due to health problems of the participant.
  Analysis only includes participants who received unpaid help (103 participants) or paid help (51 participants).
  Hours
    Unpaid help | 7.7 (10.20)
    Paid help | 2.2 (9.20)
HLQ Impediments to Work Module [Mean (Standard Deviation); unit: Units on a scale] — The HLQ impediments to paid and unpaid labor module asks participants how much they were indered by health problems at work over the past 2 weeks on a scale from not at all (0), a little (1) to very (2). Participants were also asked whether they had performed unpaid activities (household work, shopping, odd jobs/chores, childcare) according to the following: Did do, hindered (1); Did do, not hindered (0); Did not do, due to health problems (2); Did not do, due to other reasons (0). The aggregated score ranges from 0 (no impediments) to 8 (unable to do any of the surveyed activities).
  Units on a scale | 3.0 (1.33)
Physician Global Assessment [Mean (Standard Deviation); unit: Units on a scale] — The physician global assessment of disease activity asks the physician to assess how the participant is doing since their last visit on a scale from 1 (very good, asymptomatic, no limitations in normal activities) to 5 (very poor, severe symptoms that are intolerable, inability to carry out all normal activites).
  Units on a scale | 3.23 (0.463)
Patient Global Assessment [Mean (Standard Deviation); unit: Units on a scale] — The patient global assessment of disease activity is a 5-point scale concerning disease activity that asks how the participant is doing since their last visit with regard to their rheumatoid arthritis. Participants answer on a scale from 1 (very good, asymptomatic, no limitation in normal activites) to 5 (very poor, very severe symptoms that are intolerable, inability to perform all normal activites).
  Units on a scale | 3.28 (0.559)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement of ≥ 0.50 Units From Baseline to Month 24 in the HAQ DI
Description: The HAQ DI is a questionnaire which measures functional status in patients with psoriatic arthritis. The questionnaire addresses health-related quality of life issues related to psoriatic arthritis such as dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability.
Time Frame: Baseline and 24 months
Population: Full Analysis Set, composed of all participants who received at least one dose of study medication and had at least one baseline and at least one post-baseline measurement for the endpoint of interest. Imputation by last observation carried forward (LOCF) was applied.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enbrel
Number analyzed (Participants) | 109
percentage of participants | 56.0 [46.1 to 65.0]

2. Secondary Outcome: Change From Baseline to Month 24 in the Health and Labour Questionnaire (HLQ) Absence From Work Module
Description: The HLQ collects quantitative data on the relation between illness and treatment and work performance. The instrument is divided into 4 modules to collect data about absence from work, reduced productivity at paid work, unpaid labor production and impediments to paid and unpaid labor. The absence from work module asks participants to indicate how many days in the past 2 weeks they missed work due to health problems. Change from Baseline was calculated as the Baseline value - Month 24 value. A positive change from Baseline value indicates improvement.
Time Frame: Baseline and 24 months
Population: Full Analysis Set participants who completed the HLQ at Baseline and Month 24, and were employed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Enbrel
Number analyzed (Participants) | 40
days | 0.4 (2.64)

3. Secondary Outcome: Change From Baseline to Month 24 in the HLQ Reduced Productivity at Paid Work Module
Description: The HLQ collects quantitative data on the relation between illness and treatment and work performance. The instrument is divided into 4 modules to collect data about absence from work, reduced productivity at paid work, unpaid labor production and impediments to paid and unpaid labor. In the reduced productivity at work module participants were asked to estimate the number of additional hours required to compensate for production losses due to illness on working days over the past 2 weeks.
  Change from Baseline was calculated as the Baseline value - Month 24 value. A positive change from Baseline value indicates improvement.
Time Frame: Baseline and Month 24
Population: Full Analysis Set participants who completed the HLQ at Baseline and Month 24, were employed, and indicated they had some production losses due to health problems at work (participants with no production losses were not included).
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Enbrel
Number analyzed (Participants) | 2
Hours | 0.0 (0.00)

4. Secondary Outcome: Change From Baseline to Month 24 in the HLQ Unpaid Labour Production Module
Description: The HLQ collects quantitative data on the relation between illness and treatment and work performance. The instrument is divided into 4 modules to collect data about absence from work, reduced productivity at paid work, unpaid labor production and impediments to paid and unpaid labor. The Unpaid Labour Production Module assesses the amount of hours of unpaid work (including household work, shopping, caring for children and odd jobs around the house), normally performed by the participant, that were taken over by other members of the household, family or friends (unpaid help), and/or by paid workers due to health problems of the participant. Change from Baseline was calculated as the Baseline value - Month 24 value. A positive change from Baseline value indicates improvement.
Time Frame: Baseline and month 24
Population: Full Analysis Set participants who completed the HLQ at Baseline and Month 24 and who performed any unpaid work at both time points (71 participants). "n" indicates the number of participants who had unpaid or paid help with their unpaid work.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Enbrel
Number analyzed (Participants) | 71
Hours
  Unpaid help (n=66) | 3.2 (12.06)
  Paid help (n=27) | 1.9 (11.39)

5. Secondary Outcome: Change From Baseline to Month 24 in the HLQ Impediments to Paid and Unpaid Labour Module
Description: In the HLQ impediments to paid and unpaid labor module participants were asked "Were you hindered by health problems at your paid work over the past two weeks?" and answered according to the following: 'no not at all = 0', 'yes, a little = 1', 'yes, very = 2'. Participants were also asked whether they had performed 4 unpaid activities (household work, shopping, odd jobs / chores, and childcare), and answered according to the following: Did do, hindered = 1; Did do, not hindered = 0; Did not do, due to health problems = 2; Did not do, due to other reasons = 0. The aggregated score ranges from 0 (no impediments) to 8 (unable to do any of the surveyed activities). Change from Baseline was calculated as the Baseline value - Month 24 value. A positive change from Baseline value indicates improvement.
Time Frame: Baseline and month 24
Population: Full Analysis Set participants who completed the HLQ at Baseline and Month 24 and who performed any unpaid work at both time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enbrel
Number analyzed (Participants) | 71
Units on a scale | 1.5 (1.68)

6. Secondary Outcome: Change From Baseline to Month 24 in the Physician Global Assessment
Description: The physician global assessment of disease activity asks the physician to assess how the participant is doing since their last visit on a scale from 1 (very good, asymptomatic, no limitations in normal activities) to 5 (very poor, severe symptoms that are intolerable, inability to carry out all normal activites). Change from Baseline was calculated as Baseline value - Month 24 value. A positive change from Baseline indicates improvement.
Time Frame: Baseline and month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enbrel
Number analyzed (Participants) | 110
Units on a scale | 0.91 (0.991)

7. Secondary Outcome: Percent Change From Baseline to Month 24 in Physician Global Assessment
Description: The physician global assessment of disease activity asks the physician to assess how the participant is doing since their last visit on a scale from 1 (very good, asymptomatic, no limitations in normal activities) to 5 (very poor, severe symptoms that are intolerable, inability to carry out all normal activites).
  Percent change from Baseline was calculated as (Baseline value - Month 24 value) / Baseline value * 100. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Mean (Full Range); unit: Percentage change
Arm/Group | Enbrel
Number analyzed (Participants) | 110
Percentage change | 27.2 [-66.7 to 75.0]

8. Secondary Outcome: Change From Baseline to Month 24 in Patient Global Assessment
Description: The patient global assessment of disease activity is a 5-point scale that asks how the participant is doing since their last visit with regard to their rheumatoid arthritis. Participants answer on a scale from 1 (very good, asymptomatic, no limitation in normal activites) to 5 (very poor, very severe symptoms that are intolerable, inability to perform all normal activites). Change from Baseline was calculated as Baseline value - Month 24 value. A positive change from Baseline indicates improvement.
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Enbrel
Number analyzed (Participants) | 109
Units on a scale | 0.59 (0.874)

9. Secondary Outcome: Percent Change From Baseline to Month 24 in Patient Global Assessment
Description: The patient global assessment of disease activity is a 5-point scale that asks how the participant is doing since their last visit with regard to their rheumatoid arthritis. Participants answer on a scale from 1 (very good, asymptomatic, no limitation in normal activites) to 5 (very poor, very severe symptoms that are intolerable, inability to perform all normal activites). Percent change from Baseline was calculated as (Baseline value - Month 24 value) / Baseline value * 100. A positive change from Baseline indicates improvement.
Time Frame: Baseline and month 24
Population: Full Analysis Set, composed of all participants who received at least one dose of study medication and had at least one baseline and at least one post-baseline measurement for the endpoint of interest. Imputation by last observation carried forward (LOCF) was applied. Change was based on paired data.
Measure: Mean (Full Range); unit: Percentage change
Arm/Group | Enbrel
Number analyzed (Participants) | 109
Percentage change | 16.4 [-33.3 to 75.0]

10. Secondary Outcome: Percentage of Participants With Improvement of ≥ 75 Percent From Baseline to Month 24 in the Psoriasis Activity and Severity Index (PASI)
Description: The PASI was is a method for quantifying the intensity of psoriasis, and for evaluating its improvement with treatment. This index is based on the quantitative assessment of three typical signs of psoriatic lesions: erythema, infiltration, and desquamation, combined with the skin surface area involvement. The index has a range from 0.0 to 72.0, with higher scores indicating worse psoriasis.
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enbrel
Number analyzed (Participants) | 110
percentage of participants | 41.8 [32.5 to 51.6]

11. Secondary Outcome: Percentage of Participants With a Psoriatic Arthritis Response Criteria (PsARC) Response at Month 24
Description: Psoriatic Arthritis Response Criteria response is defined as improvement from Baseline in at least 2 of 4 criteria, one of which must be joint pain /tenderness or swelling and no worsening in any of the 4 following criteria: • Joint Pain/Tenderness score: Physician assessment of 78 joints for pain/tenderness on a scale from 0 (none) to 3 (severe) with a total score ranging from 0 to 234, with higher scores indicating more severe disability; • Joint Swelling score: Physician assessment of 78 joints for swelling on a scale from 0 (none) to 3 (severe) with a total score ranging from 0 to 234 with higher scores indicating more severe disability; • Patient global assessment of disease activity: Measured on a 5-point scale from 1 (very good) to 5 (very poor); • Physician global assessment of disease activity: Measured on a 5-point scale from 1 (very good) to 5 (very poor).
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enbrel
Number analyzed (Participants) | 109
percentage of participants | 78.9 [70.0 to 86.1]

ADVERSE EVENTS:
Time Frame: Up to 25 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Enbrel
Serious Adverse Events (participants affected / at risk) | 14/110
Other Adverse Events (participants affected / at risk) | 67/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (N=110)
Angina pectoris (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Appendicitis perforated (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enbrel (N=110)
Diarrhoea (Gastrointestinal disorders) | 7
Influenza like illness (General disorders) | 11
Injection site reaction (General disorders) | 13
Nasopharyngitis (Infections and infestations) | 20
Sinusitis (Infections and infestations) | 10
Upper respiratory tract infection (Infections and infestations) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Hypertension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.